CLINICAL TRIAL: NCT01242878
Title: MACS Study - Microparticles and Coagulation in Sickle Cell Disease: An Observational Study to Measure the Levels of Circulating Microvesicles and Coagulation Activation Parameters in Patients With Sickle Cell Disease in the in- and Out-patient Setting.
Brief Title: MACS Study - Microparticles and Coagulation in Sickle Cell Disease
Acronym: MACS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); The Whittington Hospital NHS Trust (Other Government)
Responsible Party: Professor John Porter, University College London
Other Study IDs: 10/0270
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Sickle Cell Disease
Keywords: HbSS; Sickle cell anemia; HbSC; HbSbetathalassemia; Hemoglobinopathy; Hemoglobinopathies
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobinopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma will be retained following appropriate informed written consent for further ethically approved studies as stipulated on the consent forms
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy volunteers: ethnically matched people who do not have sickle cell disease
- patients: sickle cell disease patients

SUMMARY:
Sickle cell disease (SCD) is an inherited disorder of the red blood cell. It is now the commonest genetic disorder in the UK and of childhood stroke, with up to 40% of children having a stroke (clinical or picked up on a scan) by school age. Patients are prone to develop acute crises necessitating hospital admission and resulting in long-term complications. Such events result in considerable morbidity, disability and mortality with its consequent burden on patients, families, the health service and society as a whole. Doctors have very little ability to predict who will get ill and when and so it is very difficult to known when and how to administer treatments. Furthermore there is very little in the way of treatments available and the mainstay of prevention is a chronic blood transfusion programme which is expensive, requires time off work and school and can be fraught with complications. This, in a population who is frequently educationally and socially disadvantaged at the outset. Recent evidence in sickle cell disease and other diseases that have similar underlying processes, points towards the importance of microparticles (circulating broken pieces of cells) and the coagulation system as being important. By comparing levels of these particles and molecules in patients with those found in healthy volunteers and with other measures known to be important, this study hopes to identify their role so as to improve the management of these patients and potentially to lead the way for new therapies. Participants will be required to donate a small amount of blood (1 teaspoon in the very young, two in older children and adults). The investigators aim to take this sample where possible when people are having a blood test in any case.

DETAILED DESCRIPTION:
Purpose and design

* Why is it needed? The purpose of this study is to try and identify a measurable parameter to act as a disease indicator in sickle cell disease. The reason such a parameter is needed is that although patients seem to have the same genetic defect, they can have enormously different outcomes ranging from mild illness to stroke, catastrophic chest disease, kidney failure and death. Currently we have no real tools to properly prognosticate. This means it is difficult to know when to intervene in an illness and when to scale down and stop treatment. The repercussions of not intervening in a timely manner can be catastrophic and it is known that children who develop stroke have future ongoing and progressive intellectual deficits. The identification of a disease indicator could have potential for therapeutic innovation in the future. This is important as much of the current treatments are blunt, expensive and not always effective. In addition there is a paucity of treatment options for the clinician and those that are available e.g. blood transfusion are expensive socially and financially, have medical complications and are realistically not available for the majority of people who have sickle cell disease.
* Why microparticles and coagulation markers? An excellent candidate for the role of disease prognosticator is coagulation markers and microparticles. Microparticles and coagulation markers have been shown by members of this investigative group to be elevated in sickle cell disease and in other paediatric vascular diseases. There has been a lot of interest in the haematology world of late in these particles with papers and presentations and all the international conferences - EHA (European Haematology Association), BSH (British Society of Haematology) and ASH (American Society of Hematology), though these have been performed on small selected groups, frequently on adults only and only rarely with any sort of controls. What has not been done so far is to compare these levels to ethnically matched people or to measure these in children with sickle cell disease. This is remiss as it is known that the vascular changes occur right from the beginning of life with children have symptoms and signs of vasculopathy often by 6 months of age and with up to 40% having had some sort of stroke by school entry. What also has been omitted is performing these tests in a larger cohort and comparing with the variety of current measures of disease severity and measure of vasculopathy. It is only with this kind of information can we make proper inferences about the importance of these measures and go on to develop studies where these are used as disease prognosticators and one day even as a target for therapeutic intervention.
* Why here and now? Here and now presents a perfect opportunity for this study. Dr Trompeter is the author of the study and will be coordinating the study. She is currently a locum Consultant Haematologist at UCLH and a Specialist Registrar in Haemoglobinopathies at Guy's and St Thomas' and has been looking after the in- and out-patients with sickle cell disease at these sites. She has also been involved in ongoing studies in sickle cell disease at these sites as an investigator. Furthermore she has worked in a similar clinical capacity at both UCLH and The Whittington Hospital and has built up a good rapport and working relationship with staff, patients and their families at these sites. She is registered for a PhD at UCL and has already performed these assays as part of the original ongoing study in adults with sickle cell disease, which has papers published and soon to be submitted. These sites in combination represent one of the largest cohort of sickle cell patients in the country. The centres have been externally audited as part of the sickle peer review and have had their considerable qualities assessed and lauded. They have the capacity, ability and habit of measuring all the other parameters of interest in this study as a matter of routine clinical care. The clinicians have enormous experience and rapport with their patients but also have a considerable research repertoire. The Professors and scientists in this study have all demonstrated their immense knowledge and expertise in the fields of sickle cell disease and vasculopathy and are internationally renown, leading many important related studies. They have provided much of the support and scientific rationale to the designing of this study. The investigators are well known to the sickle community and its representatives and the author has spoken with patients groups who persistently express a desire for medical advancement and showed a real interest and support for this study. This conglomeration of sites, clinicians, experts and patients represents the most exciting opportunity for advancing the understanding of sickle cell disease.

Recruitment

* Participants will be identified by the Investigator (who is part of their normal care team) from the in- or out-patient setting as having met the inclusion criteria. Patients with sickle cell disease attend dedicated clinics and are well known to the investigators. The consent procedures are described below. There will be no payment.
* In the case of the patients, they will then progress to have their scheduled blood test as part of their normal clinic care, onto which a further blood sample (1 teaspoon in the case of small children, 2 teaspoons in the case of older children and adults) will be obtained for the purpose of this study.
* There are two groups of healthy volunteers - adults and children. They should be ethnically matched. The majority of the adults can be identified from the sickle clinic setting as family members attending with their patient relative. These people have the additional advantage of knowing their sickle status. There are also many ethnically matched members of staff or other people attending the hospital that may want to be involved in the study. Some adult volunteers will have a blood sample for the purpose of the study only, others will be having blood tests in any case and the study sample being taken in addition, if they do not know their sickle status they will be tested. They will consent separately for this and the information given back to them regarding this second test. Separate consent will also be taken for reporting to them and their G.P. also. Ethnically matched children healthy volunteers will be identified from the in and outpatient setting. They are extremely likely to know their sickle status in any case because of the national screening programme. Children will only participate in the study if they are having a blood tests in any case.

ELIGIBILITY:
Inclusion Criteria:

* Subject Inclusion Criteria:

Patient (or parent if child) able to give informed consent Compound heterozygote or homozygote for a sickling disorder (i.e. has sickle cell disease) Having a blood test in any case

* Healthy volunteer Inclusion Criteria:

Person (or parent if child) able to give informed consent If a child, having a blood test or cannula inserted in any case Ethnically matched - of African origin Must know their sickle cell status or have it tested as part of the study and agree to have this result given to them and their G.P.

Exclusion Criteria:

* Subject Exclusion Criteria:

Inability to meet all inclusion criteria

* Healthy Volunteer Exclusion Criteria:

Compound heterozygote or homozygote for a sickling disorder (i.e. has sickle cell disease) Inability to meet all inclusion criteria Ongoing cancerous/inflammatory/haematological/infective illness (the levels of microparticles and coagulation parameters have been shown to be elevated in these disorders and so would not be appropriate to be included in a control group)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This is an observational case-control study in adults and children with sickle cell disease. The cases are any child or adult attending the study centres with a confirmed diagnosis of sickle cell disease that meet the eligibility criteria. The controls are ethnically matched volunteers who meet the appropriate eligibility criteria for controls and who do not have sickle cell disease and will be recruited from the same study sites.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2010-12

CONTACTS AND LOCATIONS:
Overall Officials: John B Porter, MB BChir FRCPath MD, Principal Investigator — University College London and University College London NHS Foundation Trust; Baba Inusa, MB BS FRCPCH, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Bernard A Davis, MD FRCPath, Principal Investigator — Whittington Hospital NHS Trust
Locations (3):
- United Kingdom (3):
  - Whittington Hospital NHS Trust, London
  - University College London Hospitals NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London